CLINICAL TRIAL: NCT03601247
Title: Efficacy of Silicone Gel Versus Placebo for Postsurgical Scars of the Eyelid
Brief Title: Silicone Gel for Postsurgical Scars of the Eyelid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2018-9074
Record Dates: First submitted 2018-07-04; First posted 2018-07-26 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Scarring Due to Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- All patients (Other): Split-face study: patients undergoing bilateral eye surgery will have the sides of their face randomized to receive either placebo or silicone gel.
  Interventions: Device: silicone gel

INTERVENTIONS:
Device: silicone gel — Patients who have consented to the study will receive two tubes labeled only "left" and "right", corresponding to the side of the face to which the tube contents will be applied. One tube will contain silicone gel and the other tube will contain aquaphor. Neither the patient nor the surgeon will know what side will receive which treatment. These tubes will be given to patients at post-operative week 1 visit. Patients will be instructed to rub the solution into their eyelid incisions gently with their fingers for 2-3 minutes twice a day

SUMMARY:
To determine whether silicone gel is effective at preventing or minimizing scar formation after eyelid surgery.

DETAILED DESCRIPTION:
Upper eyelid blepharoplasty or ptosis repair is performed when the upper eyelid becomes droopy, which often occurs as a natural part of the aging process. The droopiness of the upper eyelids decreases the ability to see objects in their peripheral vision, causing functional deficits. Additionally, the droopiness can be a cosmetic concern for many. The most effective treatment option is blepharoplasty or ptosis repair.

During routine pre-operative counseling, many patients note a fear of prominent facial scarring. Different techniques have been described in the literature to minimize scarring, from steroid creams to injections to laser therapy; however, there is currently no consensus for long-term management of post-surgical eyelid scars. Specifically, there is no study examining the efficacy of topical silicone gel on eyelid scars, although a few studies have examined its efficacy on other facial scars. Silicone is proposed to aid in healing by regulating fibroblast production, reducing collagen production, and modifying expression of growth factors.

The investigator's study is designed to determine whether topical silicone may prevent significant post-operative eyelid scar formation. It may help clarify whether there is a safe and effective topical treatment for patients undergoing eyelid surgery for whom scarring or cosmesis is a concern. It is the first study of silicone gel on the eyelid and is also prospective, randomized, and double blinded.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included if they have met the criteria for undergoing upper eyelid ptosis repair or blepharoplasty. This means they have droopiness of the upper eyelids that is visually significant and limiting the patient's visual field.

Exclusion Criteria:

* Patients will be excluded if they require additional upper eyelid surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2024-01-11 (Actual); Study Completion 2024-01-11 (Actual)

PRIMARY OUTCOMES:
The appearance of post-operative scarring as graded by a blinded third-party physician using a questionnaire | 2 years
  To determine whether silicone gel is effective at preventing or minimizing scar formation after eyelid surgery.

SECONDARY OUTCOMES:
Rates of patient satisfaction with their post-operative scars as assessed by a questionnaire | 2 years
  To determine whether silicone gel treatment has any effect on patient satisfaction with post-surgical eyelid scars.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Barmettler, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No